CLINICAL TRIAL: NCT04015076
Title: A Phase 1, Randomised, Double-Blind, Placebo Controlled, Single and Multiple Ascending Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Inzomelid in Healthy Adult Participants as Well as an Open Label Cohort to Confirm the Safety, Pharmacokinetics, and Pharmacodynamics of Inzomelid in Adult Patients With Cryopyrin-Associated Periodic Syndromes
Brief Title: Safety and Tolerability, Pharmacokinetic and Pharmacodynamic Study With Inzomelid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inflazome UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IZD174-001
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (Experimental): Inzomelid or Placebo
  Interventions: Drug: Inzomelid; Drug: Placebo
- Multiple Ascending Dose (Experimental): Inzomelid or Placebo
  Interventions: Drug: Inzomelid; Drug: Placebo
- Patients with CAPS (Experimental): Inzomelid Open Label
  Interventions: Drug: Inzomelid

INTERVENTIONS:
Drug: Inzomelid — Active Drug
Drug: Placebo — Placebo to Match
  Arms: Multiple Ascending Dose; Single Ascending Dose

SUMMARY:
This is a first in human (FIH), single-centre, double blind, randomised, cross-over, SAD followed by a MAD study of Inzomelid. The study is designed to evaluate the safety, tolerability, PK, PD, and food effect of Inzomelid in healthy adult participants and to evaluate the safety, tolerability, PK, PD, and preliminary clinical efficacy of Inzomelid in adult patients with CAPS. Oversight will be provided by a safety monitoring committee (SMC) comprised of the Investigator, the Sponsor's Medical Monitor and an Independent Medical Monitor.

ELIGIBILITY:
Inclusion Criteria- Healthy Volunteers:

* Healthy male or female volunteers, aged 18 to 65 years (inclusive at the time of informed consent);
* Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of study drug;
* Participants must have a Body Mass Index (BMI) between ≥18.0 and ≤32.0 kg/m2 at Screening;

Inclusion Criteria- CAPS Patients:

* Patients with a confirmed diagnosis of CAPS (FCAS, NOMID, or MWS) aged 18 to 70 years (inclusive at the time of informed consent);

Exclusion Criteria- Healthy Volunteers:

* Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period;
* Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant;
* Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol;

Exclusion Criteria- CAPS Patients:

* Live vaccinations within 3 months prior to Screening, for the duration of the study and for up to 3 months following the last dose of study drug;
* Positive QuantiFERON test at the Screening visit or within 2 months prior to Screening.

Participants who have a positive QuantiFERON test with documentation of BCG vaccination, who are at low environmental risk for TB infection or reactivation, and have a negative chest X-ray can be included;

* Pregnant or lactating at Screening or planning to becomepregnant (self or partner) at any time during the study, including the follow-up period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent advert events [Safety and Tolerability] | Day 1-8 for SAD, Day 1-16 for MAD
  Incidence, frequency and severity of treatment emergent advert events
Peak Plasma Concentration (Cmax)-single dose | Day 1-3
  Peak plasma concentration following single dose administration
Area under the plasma concentration versus time curve (AUC)- single dose | Day 1-3
  AUC following single dose administration
Peak Plasma Concentration (Cmax)-multiple dose | Days 1-9
  Peak plasma concentration following multiple dose administration
Area under the plasma concentration versus time curve (AUC)- multiple dose | Days 1-9
  AUC following multiple dose administration
Peak Plasma Concentration (Cmax)-multiple dose | Days 1-16
  Peak plasma concentration following multiple dose administration
Area under the plasma concentration versus time curve (AUC)- multiple dose | Days 1-16
  AUC following multiple dose administration

SECONDARY OUTCOMES:
Pharmacodynamic activity | Day 1-3 for SAD and Day 1-9 for MAD
  NLRP3 Inhibition in whole blood
Reduction in CAPS symptom scores | Days 1-15
  Reduction in Physician Assessed CAPS scores based on 8 point questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ben Snyder, MB, BS, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Melbourne, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No